CLINICAL TRIAL: NCT07349836
Title: Application of mRNA Immunotherapy Technology in EB Virus Related Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Xi Zhang, MD, Professor, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNP-mRNA for EBV
Record Dates: First submitted 2026-01-02; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: EBV-associated Tumors
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WGc-043 Injection, monotherapy (Experimental)
  Interventions: Biological: WGc-043 injection
- WGc-043 injection, combination therapy (Experimental)
  Interventions: Biological: WGc-043 injection; Biological: Immune Checkpoint Inhibitors; Drug: Standard therapy

INTERVENTIONS:
Biological: WGc-043 injection — WGc-043 injection
Biological: Immune Checkpoint Inhibitors — Immune checkpoint inhibitors
  Arms: WGc-043 injection, combination therapy
Drug: Standard therapy — Standard therapy
  Arms: WGc-043 injection, combination therapy

SUMMARY:
EB virus is associated with various epithelial and lymphoid derived tumors, such as Burkitt lymphoma, Hodgkin lymphoma, epithelial derived nasopharyngeal carcinoma, and some gastric cancers. In EBV related tumors, epithelial tumors account for over 80%, with the majority being nasopharyngeal carcinoma and EVB related gastric cancer. Among lymphomas, NK/T-cell lymphoma is the lymphoma most closely associated with EBV infection, accounting for approximately 6%. In the world, the incidence rate of NK/T lymphoma in China is the highest, and it is a malignant lymphoma with rapid development and strong invasion.

mRNA immunotherapy is a promising novel anti-tumor treatment method. Previous basic research and clinical practice have shown that immune drugs prepared using antigen-presenting cells loaded with tumor antigens, CAR-T cells, etc. can produce objective clinical therapeutic effects. Compared with traditional immune drugs, mRNA immune drugs have unique advantages in the field of tumor immunotherapy. They can express and present antigens for a long time, thereby stimulating stronger immune responses and producing cytotoxic T cells (CTLs) that specifically recognize EB virus antigens, exerting anti-tumor effects.

Previous studies have preliminarily confirmed that the mRNA immunotherapy monotherapy has good safety and tolerability in various tumor populations. Considering that most EBV positive tumor patients have limited treatment options, and that PD-1/L1 inhibitors have shown excellent anti-tumor efficacy in the treatment of various malignant tumors, research on mRNA vaccine monotherapy and its combination with immune checkpoint inhibitors is being conducted to provide more treatment options for patients with EB virus related tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients aged ≥ 18 years old;
* 2. Diagnosed with EBV related diseases through histology or cytology, including but not limited to nasopharyngeal carcinoma, gastric cancer, lymphoma, EBV disease after HSCT etc;
* 3. ECOG physical condition score: 0-2 points;
* 4. Expected survival period ≥ 3 months;
* 5. The main organ functions well, that is, the relevant examination indicators meet the requirements;
* 6. The subject has no pregnancy plan during the treatment period and agrees to voluntarily take effective contraceptive measures during the trial period and within 4 months of stopping treatment, and the pregnancy of women of childbearing age is negative;
* 7. Able to understand and voluntarily sign a written informed consent form before the experiment;
* 8. Able to communicate well with researchers and complete experiments according to the protocol.

Exclusion Criteria:

* 1. The patient has a history of other tumors in the past, except for the cured skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, gastrointestinal intramucosal carcinoma and other malignant tumors that the researchers think can be included;
* 2. Central nervous system (CNS) tumors or CNS metastases;
* 3. Chest fluid, ascites, and pericardial effusion that require drainage due to clinical symptoms; Hepatic encephalopathy, hepatorenal syndrome, or Child Pugh B or more severe cirrhosis;
* 4. Known to have invasive NK cell leukemia or NK lymphoblastic leukemia/lymphoma; Or accompanied by hemophilic cell syndrome;
* 5. There are any uncontrollable clinical or mental illnesses or other major illnesses that, according to the researcher's assessment, may hinder the provision of informed consent, interfere with the interpretation of the trial results, pose risks to the subjects participating in this trial, or otherwise affect the achievement of the trial objectives;
* 6. Allergic to the experimental drug (including any excipients). Previous history of severe allergies to any medication, food, or vaccine, such as anaphylactic shock, allergic laryngeal edema, allergic dyspnea, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc;
* 7. The most recent anti-tumor treatment (radiotherapy, chemotherapy, targeted therapy, immunotherapy, or local regional therapy) is less than 4 weeks after the first dose or within 5 half lives of the drug (whichever is shorter), or palliative radiotherapy is less than 2 weeks after the first dose; Patients with adverse reactions related to anti-tumor therapy (excluding hair loss) that have not recovered to NCI CTCAE ≤ 1 or inclusion criteria after previous anti-tumor therapy;
* 8. Subjects who receive systemic therapy with corticosteroids (>10 mg/day of prednisone or equivalent doses of other corticosteroids) or other immunosuppressive agents within 14 days prior to their first administration. In the absence of active autoimmune diseases, inhalation or topical use of steroids and adrenal hormone replacement with a dose ≤ 10 mg/day of prednisone efficacy dose is allowed;
* 9. Within 6 months prior to the first administration, have received mRNA vaccines or lipid nanoparticles (LNP) equivalent nanoparticles for drug delivery;
* 10. Having undergone major surgery within the 4 weeks prior to screening (excluding minor surgeries such as catheter insertion or biopsy surgery as required by the protocol), or the impact of surgery or trauma has been eliminated for less than 14 days prior to enrollment;
* 11. Have a history of drug abuse or known medical, psychological, or social conditions, such as a history of alcohol or drug abuse;
* 12. Known active infections such as hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), syphilis, etc.:
* 13. The researchers believe that there are any other factors that are not suitable for the subjects to enter this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: incidence and severity of adverse effects | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 2 years
Disease control rate (DCR) | Through study completion, an average of 2 years
Progression free survival (PFS) | From date of initial treatment until the date of first comfired progression or date of death from any cause, whichever came first, assessed up to 24 months